CLINICAL TRIAL: NCT04857658
Title: Effect of Extraction Versus Non-extraction Orthodontic Treatment on the Third Molars: A Non-Randomized Clinical Trial /a Prospective Clinical Trial
Brief Title: Effect of Extraction Versus Non-extraction Orthodontic Treatment on the Third Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Aboalnaga, amira ahmed aboalnaga, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEBD-CU-2021-10-4
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Orthodontic Treatment Via Premolar Extraction
Keywords: third molar impaction, third molar angulation, third molar vertical position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extraction treatment (Active Comparator): patients will be referred for extraction of the upper and lower first premolars to relieve the crowding.
  Interventions: Procedure: extraction orthodontic treatment plan
- non-extraction treatment (No Intervention): Leveling and alignment of the moderate crowding will be performed through a recall visits of 4 weeks for wire activation. inter-proximal reduction step might be done if needed.

INTERVENTIONS:
Procedure: extraction orthodontic treatment plan — patients will be referred for extraction of the upper and lower first premolars then orthodontic treatment will follow.
  Arms: extraction treatment

SUMMARY:
What is the effect of extraction orthodontic treatment in comparison to non- extraction treatment on the position, inclination and incidence of impaction of the third molars?

DETAILED DESCRIPTION:
Data regarding the personal information (name, age and gender), chief complaint, medical and dental history will be taken. Medical history questionnaire will be filled by the patient to exclude the presence of any systemic conditions.

complete set of orthodontic records will be taken; Pre- operative records including (standardized intra- and extra-oral photographs, primary impression for study model, panoramic & lateral cephalogram). After formulating the best treatment plan for each patient, All patients will be enrolled into one of two groups: Intervention Group (I) : Extraction treatment group. Comparator group (C): Non-extraction group. Following the end of treatment, Post-treatment records including (standardized intra- and extra-oral photographs, primary impression for study model, panoramic & lateral cephalogram) will be taken.

Primary outcome: The angulation of the mandibular third molars.Secondary outcomes:

1. space available for the upper and lower third molar.
2. Angulation of the third molar.
3. The vertical position of the third molars.
4. the mineralization status of the third molars

ELIGIBILITY:
Inclusion Criteria:

* Adolescent males and females (14-18 years) with Bilaterally unerupted developing third molars. Not more than two thirds of the root development of the third molars had taken place.

  * Dental Class I malocclusion cases requiring four premolar extraction with a moderate anchorage requirement.
  * low or increased vertical dimension.

Exclusion Criteria:

* Premolar extraction cases requiring maximum anchorage preparation.

  * Low vertical dimension.
  * patients without dentofacial deformities, severe facial asymmetries, or missing teeth.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
third molar angulation | at the end of orthodontic treatment
  The angulation of the mandibular third molars

SECONDARY OUTCOMES:
space available for the upper and lower third molar | at the end of orthodontic treatment
  space available for the upper and lower third molar
Angulation of the third molar. | at the end of orthodontic treatment
  Angulation of the third molar.
The vertical position of the third molars | at the end of orthodontic treatment
  The vertical position of the third molars
the mineralization status of the third molars | at the end of orthodontic treatment
  the mineralization status of the third molars

CONTACTS AND LOCATIONS:
Overall Officials: amira aboalnaga, Principal Investigator — Cairo University
Locations (1):
- Amira Aboalnaga, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
the pre-treatment and post-treatment records